CLINICAL TRIAL: NCT02745067
Title: Effectiveness of Enhanced Cognitive Behavioral Therapy (CBT-E) in the Treatment of Anorexia Nervosa: a Prospective Multidisciplinary Study
Brief Title: Effectiveness of Enhanced Cognitive Behavioral Therapy (CBT-E) in the Treatment of Anorexia Nervosa
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Haukeland University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2015/2328
Record Dates: First submitted 2016-04-13; First posted 2016-04-20 (Estimated); Last update posted 2025-03-26 (Actual); Status verified 2022-03

CONDITIONS: Anorexia Nervosa
MeSH Terms: conditions — Anorexia Nervosa

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Enhanced cognitive behavioral therapy (Other): Enhanced cognitive behavioral therapy (CBT-E) for eating disorders
  Interventions: Behavioral: enhanced cognitive behavioral therapy

INTERVENTIONS:
Behavioral: enhanced cognitive behavioral therapy

SUMMARY:
The primary objective of this study is to gain knowledge about the effectiveness of enhanced cognitive behavioral therapy (CBT-E) for anorexia nervosa (AN).

DETAILED DESCRIPTION:
The study will assess the potency of outpatient CBT-E in a sample of patients suffering from AN who are admitted to the Section for Eating Disorders at the Department for Psychosomatic Medicine, Haukeland University Hospital in Bergen, Norway.

Secondary objectives are to (1) prospectively identify baseline predictors of treatment outcome and dropout, (2) determine variables related to the treatment process and patient engagement as predictors of the outcome and/or treatment dropout, and (3) in a multidisciplinary approach, focus on selected pathophysiological mechanisms including changes in the gut microbiota as well as immunological measures in patients with severe AN in different stages of the disease, and determine to what extent they are related to treatment outcome.

ELIGIBILITY:
Inclusion Criteria:

* patients aged >16 years
* suffering from AN, as diagnosed based on the Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition (DSM-V) and confirmed with a clinical examination.
* either at least one unsuccessful treatment attempt in a secondary health-care service unit or severe AN that is evaluated as not manageable in a secondary health-care service unit.

Exclusion Criteria:

* deemed unsafe to manage on an outpatient basis
* psychiatric comorbidity that precludes a focused eating-disorder treatment, such as psychosis or drug abuse.
* not available to participate during the requested treatment period
* for the analysis of the gut microbiota: patients suffering from inflammatory bowel disease, acute or chronic diarrhea or other bowel disease, treatment with antibiotics during the previous 3 months before stool sampling, or laxative abuse;

Min Age: 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2016-09 (Actual); Primary Completion 2021-12 (Actual); Study Completion 2022-01 (Actual)

PRIMARY OUTCOMES:
Eating Disorder Examination Questionnaire (EDE-Q), score | 1 year
BMI | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Ute Kessler, PhD, Principal Investigator — Haukeland University Hospital
Locations (1):
- Haukeland University Hospital, Bergen, Norway

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Kessler U, Kleppe MM, Rekkedal GA, Ro O, Danielsen Y. Experiences when implementing enhanced cognitive behavioral therapy as a standard treatment for anorexia nervosa in outpatients at a public specialized eating-disorder treatment unit. J Eat Disord. 2022 Feb 5;10(1):15. doi: 10.1186/s40337-022-00536-7. PMID 35123583
- [Derived] Kleppe MM, Kessler U, Rekkedal GA, Skjakodegard HF, Danielsen YS. Differences in sleep patterns between patients with anorexia nervosa and healthy controls: a cross-sectional study. J Eat Disord. 2023 May 16;11(1):76. doi: 10.1186/s40337-023-00799-8. PMID 37194104
- [Derived] Kleppe MM, Bronstad I, Lied GA, Danielsen Y, Rekkedal GA, Kessler U. Intestinal barrier integrity in anorexia nervosa (a pilot study). Int J Eat Disord. 2022 May;55(5):703-708. doi: 10.1002/eat.23678. Epub 2022 Jan 17. PMID 35040160
- [Derived] Kessler U, Rekkedal GA, Ro O, Berentsen B, Steinsvik EK, Lied GA, Danielsen Y. Association between gastrointestinal complaints and psychopathology in patients with anorexia nervosa. Int J Eat Disord. 2020 May;53(5):532-536. doi: 10.1002/eat.23243. Epub 2020 Feb 10. PMID 32040232
- [Derived] Danielsen YS, Ardal Rekkedal G, Frostad S, Kessler U. Effectiveness of enhanced cognitive behavioral therapy (CBT-E) in the treatment of anorexia nervosa: a prospective multidisciplinary study. BMC Psychiatry. 2016 Oct 5;16(1):342. doi: 10.1186/s12888-016-1056-6. PMID 27716162